CLINICAL TRIAL: NCT05090449
Title: No Pharmacokinetic Interaction Between Chlorthalidone and Losartan, in Healthy Volunteers Under Fasting Conditions, Administered in Fixed Combination Against Individual Components Administered Jointly and Separately
Brief Title: Non-interaction Study of Chlorthalidone and Losartan in Fixed Combination, in Healthy Subjects, Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CLRLSR-32-SIL
Record Dates: First submitted 2021-10-08; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Healthy
Keywords: Chlorthalidone; Losartan; No-interaction, pharmacokinetics; Fixed-dose combination (FDC)
MeSH Terms: interventions — Chlorthalidone; Chlorpheniramine; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A1: Individual formulation of chlorthalidone (Active Comparator): (Higroton 50, product of Sandoz, S.A. de C.V.)
  Interventions: Drug: Chlorthalidone (HIGROTON® 50)
- A2:Individual formulation Losartan (Active Comparator): (COZAAR, product of Schering Plough, S.A. de C.V., S.A. de C.V.)
  Interventions: Drug: Losartan (COZZAR®)
- A3: Co-administration of individual formulations (Active Comparator): Co-administration of individual formulations of chlorthalidone and losartan potassium
  Interventions: Drug: A1+ A2 Co-administration of Chlorthalidone and Losartan
- B: Fixed combination of chlorthalidone and losartan potassium (Experimental): B: Fixed combination of chlorthalidone and losartan potassium (product of Laboratorios Silanes S.A. de C.V.)
  Interventions: Drug: Chlorthalidone + Losartan Fixed-Dose combination

INTERVENTIONS:
Drug: Chlorthalidone (HIGROTON® 50) — Tablets with 50mg of Chlorthalidone, product de Sandoz, S.A. de C.V.
  Other Names: Chlo
  Arms: A1: Individual formulation of chlorthalidone
Drug: Losartan (COZZAR®) — Losartan potassium 100 mg tablet, a product of Schering-Plough, S.A. C.V.
  Other Names: Los
  Arms: A2:Individual formulation Losartan
Drug: A1+ A2 Co-administration of Chlorthalidone and Losartan — 50mg chlorthalidone + 100 mg losartan potassium
  Other Names: Chlo + Los
  Arms: A3: Co-administration of individual formulations
Drug: Chlorthalidone + Losartan Fixed-Dose combination — Tablets with fixed combination of Chlorthalidone 25 mg and Losartan Potassium
  Other Names: FDC
  Arms: B: Fixed combination of chlorthalidone and losartan potassium

SUMMARY:
Monocentric study of no pharmacokinetic interaction between chlorthalidone and losartan, with an open, randomized, single-dose design with four periods, four sequences and crossover in healthy volunteers, under fasting conditions, administered in fixed combination (Test product of Laboratorios Silanes, SA de CV) against the individual components administered jointly and separately (Higroton® 50, a product of Sandoz, SA de CV and Cozaar® , a product of Schering-Plow, SA de CV)

DETAILED DESCRIPTION:
The study was designed to recruit 36 healthy subjects, which were randomized for this study contemplating losses. All the volunteers whose data allowed at least one comparison to be made were included in the corresponding statistical analysis. The objective was to statistically compare the bioavailability of chlorthalidone (at normalized dose) and losartan potassium, in a non-interaction pharmacokinetic study after single-dose oral administration of a product with the fixed combination of active ingredients with respect to the individual components administered together and separately in healthy fasting volunteers. As a secondary objective, the tolerability of the presentations was evaluated based on the registry of adverse events at the end of the four study periods.

ELIGIBILITY:
Inclusion Criteria:

* The participation of the subjects was voluntarily in accordance with the guidelines proposed in the General Health Law and their consent will be obtained according to the aforementioned law. Likewise, the standards set by the Declaration of Helsinki, the Brazilian Review and Good Clinical Practices will be maintained.
* Only healthy male volunteers between 18 and 55 years of age were included. - The body mass index of the subjects should be between 18.0-27.0 kg / m2 according to Quetelet.
* The volunteers must be healthy, a criterion determined by the results of a complete medical history carried out by the doctors of the Clinical Research site and the laboratory and clinical test (12-lead electrocardiogram) carried out by a certified Clinical Laboratory and / or staff of the Center.
* The limits of variation allowed within normality in the screening visit was: blood pressure (sitting) from 90 to 129 mm Hg systolic and 60 to 79 mm Hg diastolic, heart rate between 50 and 100 beats per minute and respiratory rate between 14 and 20 breaths per minute according to current SOP with code CLI-DES-008 "Measurement of Vital Signs". Vital signs will be taken after 5 minutes of resting in a sitting position.
* Subjects willing to practice abstinence as a lifestyle or use of two family planning methods (including barrier methods, non-hormonal intrauterine device or bilateral tubal obstruction, and hysterectomy) during the course of the clinical study and up to 30 days after the last dose.
* The laboratory and test examinations that will be carried out for the inclusion of the subjects during the selection visit to the study will be:

  1. Complete hematic biometry with differential count: leukocytes, erythrocytes, hemoglobin, hematocrit, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, distribution width of erythrocytes, platelets, neutrophils, lymphocytes, monocytes, eosinophils, basophils.
  2. 27-element blood chemistry: glucose, urea, BUN, creatinine, BUN / creatinine ratio, uric acid, cholesterol, HDL cholesterol, triglyperides, LDL cholesterol, Non-HDL cholesterol, atherogenic index, total proteins, albumin, globulins, A / ratio G, total bilirubin, direct bilirubin, indirect bilirubin, ALT (alanine aminotransferase), AST (aspartate aminotransferase), alkaline phostatase, gamma-glutamyltraspeptidase, LDH, iron, calcium, sodium, potassium, and chlorine.
  3. General urine test. Physical examination (color, appearance, density); chemical examination (pH, leukocytes, nitrites, proteins, glucose, ketones, bilirubin, urobilinogen, hemoglobin); microscopic examination (leukocytes, erythrocytes, dysmorphic erythrocytes, casts, crystals, pavement cells, renal tubular cells, mucoid networks, bacteria, yeast).
  4. Hepatitis B and C serum tests: HBV surface antigen and anti-HCV Antibody.
  5. HIV serum tests: Anti-HIV [Human immunodeficiency virus] 1 and 2 antibodies.
  6. VDRL [Venereal Disease Research Laboratory] serum test.
  7. Urine drug abuse tests (qualitative) at screening visit and approximately 12 hours prior to each drug administration.
  8. Inline alcohol detection test approximately 12 hours before each drug administration.
  9. 12-lead electrocardiogram, which will be taken after 5 minutes of rest in the upright position.

Exclusion Criteria:

* Volunteers with a history of cardiovascular, kidney, liver, lung, muscle, metabolic, gastrointestinal, neurological, endocrine, hematopoietic, mental illness or other organic abnormalities. As well as those who have had a muscle trauma within the 21 days prior to the start of the study.
* Volunteers requiring any medication during the course of the study, other than the medication being studied. - Volunteers with a history of dyspepsia, gastritis, esophagitis, duodenal or gastric ulcer. - Volunteers who have been exposed to drugs known as liver enzyme inducers or inhibitors or who have taken potentially toxic drugs within the 30 days prior to the start of the study.
* Volunteers who have received any medication, including vitamins (with or without a prescription) or herbal remedies 30 days (or 7 half-lives) prior to the start of the study. - Clinically significant abnormalities in the electrocardiographic trace. - Electrolyte disturbances: hypokalemia, hyponatremia, hypercalcemia, and symptomatic hyperuricemia.
* Volunteers who have been hospitalized for any problem during the six months prior to the start of the study.
* Subjects who received investigational drugs within 90 days (3 months) prior to the study. - Subjects allergic to study drugs: chlorthalidone and sulphonamide derivatives, as well as losartan.
* Subjects who have ingested alcohol and / or carbonated beverages and / or containing xanthines (coffee, tea, cocoa, chocolate, mate, cola soft drinks) or who have ingested charcoal-grilled food or grapefruit juice within the previous 10 hours at the beginning of each hospitalization period or subjects who smoked tobacco within 10 hours prior to the start of the study.
* Subjects who have donated or lost 450 mL or more of blood within the 60 days prior to the start of the study.
* Subjects with a history of drug abuse and / or alcoholism.
* Volunteers who require a special diet for any reason or are on a different diet, for example vegetarian.
* Incapacity of any kind that makes it impossible for the volunteer to understand the nature, objective and possible consequences of the study.
* Evidence of non-cooperative attitude during the development of the study.
* Volunteers with positive urine drug abuse test or breath alcohol test.
* Volunteers who are not registered on the COFEPRIS page.
* Relationship of subordination between research subjects and researchers.
* Employees of the Sponsor and / or IFaB.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration following the treatment (Cmax) | Baseline, 0.333, 0.750, 1.000, 1.250, 1.750, 2.000, 3.000, 4.500, 5.000, 5.500, 6.000, 6.500, 7.000, 8.000, 10.000, 12.000, 18.000, 24.000, 48.000, 72.000, 96.000, 120.000 y 144.000 hours.
  Evaluate the fixed dose pharmacokinetics profile of Dexketoprofen-Vitamin B, employing the maximum observed concentration following the treatment (Cmax).
The area under the curve from time zero to the last measurable concentration (AUC 0-t) | Baseline, 0.333, 0.750, 1.000, 1.250, 1.750, 2.000, 3.000, 4.500, 5.000, 5.500, 6.000, 6.500, 7.000, 8.000, 10.000, 12.000, 18.000, 24.000, 48.000, 72.000, 96.000, 120.000 y 144.000 hours.
  Evaluate the fixed dose pharmacokinetics profile of Dexketoprofen-Vitamin B, employing the area under the curve from time zero to the last measurable concentration (AUC 0-t)using the linear trapezoidal method.
The area under the curve from time zero to infinity calculated (AUC 0-inf) | Baseline, 0.333, 0.750, 1.000, 1.250, 1.750, 2.000, 3.000, 4.500, 5.000, 5.500, 6.000, 6.500, 7.000, 8.000, 10.000, 12.000, 18.000, 24.000, 48.000, 72.000, 96.000, 120.000 y 144.000 hours.
  Evaluate the fixed dose pharmacokinetics profile of Dexketoprofen-Vitamin B, employing the area under the curve from time zero to infinity calculated (AUC 0-inf).
Time of the maximum measured concentration (Tmax) | Baseline, 0.333, 0.750, 1.000, 1.250, 1.750, 2.000, 3.000, 4.500, 5.000, 5.500, 6.000, 6.500, 7.000, 8.000, 10.000, 12.000, 18.000, 24.000, 48.000, 72.000, 96.000, 120.000 y 144.000 hours.
  Evaluate the fixed dose pharmacokinetics profile of Dexketoprofen-Vitamin B, employing time of the maximum measured concentration (Tmax).
Elimination rate (Ke) | Baseline, 0.333, 0.750, 1.000, 1.250, 1.750, 2.000, 3.000, 4.500, 5.000, 5.500, 6.000, 6.500, 7.000, 8.000, 10.000, 12.000, 18.000, 24.000, 48.000, 72.000, 96.000, 120.000 y 144.000 hours.
  Evaluate the fixed dose pharmacokinetics profile of Dexketoprofen-Vitamin B, employing the elimination rate (Ke), calculated by log-linear regression of the final phase of elimination.

SECONDARY OUTCOMES:
Registry of adverse events of the presentations [Tolerability] | 67 days
  Determined the tolerability of the presentations based on the registry of adverse events at the end of the four study periods.

CONTACTS AND LOCATIONS:
Overall Officials: Araceli G Medina Nolasco, M.D, Principal Investigator — Investigación Farmacológica y Biofarmacéutica, S.A.P.I. de C.V.; Liz J Medina Reyes, M.D, Principal Investigator — Investigación Farmacológica y Biofarmacéutica, S.A.P.I. de C.V.
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bienert A, Brzeziniski R, Szalek E, Dubai V, Grzeskowiak E, Dyderski S, Drobnik L, Wolc A, Olejniczak-Rabinek M. Bioequivalence study of two losartan formulations administered orally in healthy male volunteers. Arzneimittelforschung. 2006;56(11):723-8. doi: 10.1055/s-0031-1296781. PMID 17220048
- [Background] Das AK, Dhanure S, Savalia AK, Nayak SK, Tripathy SK. Human bioequivalence evaluation of two losartan potassium tablets under fasting conditions. Indian J Pharm Sci. 2015 Mar-Apr;77(2):190-5. doi: 10.4103/0250-474x.156583. PMID 26009652
- [Background] del Castillo D, Campistol JM, Guirado L, Capdevilla L, Martinez JG, Pereira P, Bravo J, Perez R. Efficacy and safety of losartan in the treatment of hypertension in renal transplant recipients. Kidney Int Suppl. 1998 Dec;68:S135-9. doi: 10.1046/j.1523-1755.1998.06827.x. PMID 9839298
- [Background] Dudkowski C, Karim A, Munsaka M. Effects of Food Intake on the Pharmacokinetics of Azilsartan Medoxomil and Chlorthalidone Alone and in Fixed-Dose Combination in Healthy Adults. Clin Pharmacol Drug Dev. 2016 Sep;5(5):393-8. doi: 10.1002/cpdd.249. Epub 2016 Mar 4. PMID 27514506
- [Background] Mann R, Mackay F, Pearce G, Freemantle S, Wilton L. Losartan: a study of pharmacovigilance data on 14,522 patients. J Hum Hypertens. 1999 Aug;13(8):551-7. doi: 10.1038/sj.jhh.1000880. PMID 10455478
- [Background] Pentikis HS, Henderson JD, Tran NL, Ludden TM. Bioequivalence: individual and population compartmental modeling compared to the noncompartmental approach. Pharm Res. 1996 Jul;13(7):1116-21. doi: 10.1023/a:1016083429903. PMID 8842055
- [Background] Potvin D, DiLiberti CE, Hauck WW, Parr AF, Schuirmann DJ, Smith RA. Sequential design approaches for bioequivalence studies with crossover designs. Pharm Stat. 2008 Oct-Dec;7(4):245-62. doi: 10.1002/pst.294. PMID 17710740
- [Background] Shah JV, Patel DP, Shah PA, Sanyal M, Shrivastav PS. Simultaneous quantification of atenolol and chlorthalidone in human plasma by ultra-performance liquid chromatography-tandem mass spectrometry. Biomed Chromatogr. 2016 Feb;30(2):208-16. doi: 10.1002/bmc.3537. Epub 2015 Jul 7. PMID 26096961
- [Background] Zandbergen AA, Baggen MG, Lamberts SW, Bootsma AH, de Zeeuw D, Ouwendijk RJ. Effect of losartan on microalbuminuria in normotensive patients with type 2 diabetes mellitus. A randomized clinical trial. Ann Intern Med. 2003 Jul 15;139(2):90-6. doi: 10.7326/0003-4819-139-2-200307150-00008. PMID 12859158